CLINICAL TRIAL: NCT00709657
Title: The Effect of a Single Intravitreal Anti-VEGF Therapy on Optic Nerve Head Perfusion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv. - Doz. Dr, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-060707
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Macular Degeneration; Regional Blood Flow; Vascular Endothelial Growth Factor
Keywords: Age-related macular degeneration; anti-VEGF
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; Bevacizumab; pegaptanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): patients with age-related macular degeneration, which are already scheduled for intravitreal anti-VEGF therapy in one eye are measured before and after treatment.
  Interventions: Drug: ranibizumab, bevacizumab or pegaptanib

INTERVENTIONS:
Drug: ranibizumab, bevacizumab or pegaptanib — measurements are performed one week before and after anti-VEGF intravitreal injection

SUMMARY:
Age related macula degeneration is one of the most common sight threatening diseases of the elderly. The so called wet form of AMD is caused by choroidal neovascularisation (CNV) of pathological vessels, which lead to leakage, bleeding and macular edema. Several lines of evidence suggest that vascular endothelial growth factor (VEGF) plays a key role in the induction CNV. Recent evidence indicates that overexpression of VEGF in the retinal pigment epithelium may lead to the development of CNV in experimental models, and intravitreal injection of a VEGF blocker prevents the development of experimental CNV. This hypothesis is also supported by the promising effects of anti-VEGF treatment in patients with choroidal neovascularisation. The substances currently in clinical use include ranibizumab (Lucentis®), bevacizumab (Avastin®) and pegaptanib (Macugen®).

However, from a physiological point of view, VEGF also serves as a survival factor for existing vessels and for neuronal cells. Moreover, it has been reported that VEGF induces vasodilatation, most probably by an increased production of nitric oxide. Accordingly one may hypothesize that anti-VEGF treatment is associated with ocular vasoconstriction with unknown long term results. Thus, in the current study, the investigators set out to investigate whether the ocular perfusion is affected by a single intravitreal anti-VEGF.

ELIGIBILITY:
Inclusion Criteria:

* 40 subjects ≥ 50 years of age
* Subjects with all angiographic subtypes of neovascular wet AMD, already scheduled for intravitreal anti-VEGF therapy in one eye
* Good central or eccentric fixation

Exclusion Criteria:

* History or previous Anti-VEGF therapy
* History or previous intravitreal injection with any drug
* Intraocular pressure ≥ 25
* Glaucoma
* History or presence of thromboembolic events
* Diabetes mellitus
* Blood donation during the previous 3 weeks
* Ametropy ≥ 6 dpt

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-03; Primary Completion 2010-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Optic nerve head blood flow | before, one week after and three weeks after intravitreal injection with an anti-VEGF drug

SECONDARY OUTCOMES:
Choroidal blood flow | before, one week after and three weeks after intravitreal injection with an anti-VEGF drug
Retrobulbar blood flow | before, one week after and three weeks after intravitreal injection with an anti-VEGF drug
Intraocular pressure | before, one week after and three weeks after intravitreal injection with an anti-VEGF drug
Systemic blood pressure | before, one week after and three weeks after intravitreal injection with an anti-VEGF drug

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, MD, Principal Investigator — Depatement of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria